CLINICAL TRIAL: NCT04949412
Title: Assessment of Serum Vitamin D Level in COVID-19 Infected Patients
Brief Title: Assessment of Vitamin D Level in COVID-19
Acronym: COVID19
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mona Mohammed Abdelrhman, Mona Mohammed Abdelrhman, Sohag University
Other Study IDs: Soh-Med-21-06-30
Record Dates: First submitted 2021-06-30; First posted 2021-07-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Covid19
Keywords: vitamin D; COVID-19; Severity
MeSH Terms: conditions — COVID-19 | interventions — Vitamin D Response Element

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — serum sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-severe COVID19: Patients with mild symptoms (i.e., fever, cough, expectoration, and other upper respiratory tract symptoms), and without abnormalities, or with mild changes on chest radiography, were classified as non-severe types or A mild change in chest radiography is defined by multiple small patchy shadows and interstitial changes, mainly in the outer zone of the lung and under the pleura.
  Interventions: Diagnostic Test: Vitamin D
- Severe Covid19: Severe pneumonia was defined by the presence of any of the following conditions: i) significantly increased respiration rate (RR): RR ≥30 times/minute; ii) hypoxia: oxygen saturation (resting state) ≤93%; iii) blood gas analysis: partial pressure of oxygen/fraction of inspired oxygen (PaO2) /FiO2) ≤ 300 mmHg (millimeters of Mercury); or iv) the occurrence of respiratory or other organ failure that require Intensive care unit (ICU) monitoring and treatment, or shock
  Interventions: Diagnostic Test: Vitamin D

INTERVENTIONS:
Diagnostic Test: Vitamin D — serum vitamin D level

SUMMARY:
his a prospective observational study will be conducted on 100 patients who were diagnosed as SARS-CoV2 positive. The data will be collected from isolation hospital in Sohag governorate during the period from the start of June 2021 to the end of July 2021. Patients will be followed up for at least one month to evaluate the prognosis.

DETAILED DESCRIPTION:
This a prospective observational study will be conducted on 100 patients who were diagnosed as SARS-CoV2 positive. The data will be collected from isolation hospital in Sohag governorate during the period from the start of June 2021 to the end of July 2021. Patients will be followed up for at least one month to evaluate the prognosis.

Inclusion criteria:

Patients with SARS-CoV2 positive PCR.

Exclusion Criteria:

Patients with chronic obstructive lung disease Chronic renal failure Patients with malabsorption Organ transplant recipient Pregnant women The study protocol will be approved by the scientific Research Ethical committee, Faculty of Medicine, Sohag University.

The Data will be collected after taken informed written consent from the patients:

Data about clinical manifestation including as fever, cough, dyspnea, fatigue and diarrhea.

Laboratory investigation:

CBC , liver function tests, CRP, D-dimer Serum creatinine, Random blood sugar, Serum ferritin and zwsVitamin D level

Assessment the severity of the disease:

Patients were classified into severe or mild cases based on results from chest radiography, clinical examination, and symptoms.

Patients with mild symptoms (i.e., fever, cough, expectoration, and other upper respiratory tract symptoms), and without abnormalities, or with mild changes on chest radiography, were classified as non-severe types. A mild change in chest radiography is defined by multiple small patchy shadows and interstitial changes, mainly in the outer zone of the lung and under the pleura.

Severe pneumonia was defined by the presence of any of the following conditions: i) significantly increased respiration rate (RR): RR ≥30 times/minute; ii) hypoxia: oxygen saturation (resting state) ≤93%; iii) blood gas analysis: partial pressure of oxygen/fraction of inspired oxygen (PaO2) /FiO2) ≤ 300 mmHg (millimeters of Mercury); or iv) the occurrence of respiratory or other organ failure that require Intensive care unit (ICU) monitoring and treatment, or shock 6.

Statistical analysis:

Continuous variables were expressed as mean ± standard deviation or median and interquartile range and compared with the student's t-test or Mann-Whitney U test according to the distribution of data. Categorical variables were presented as numbers and percentages and compared using the chi squared test or the Fisher exact test as appropriate. Spearman P rho was used to assess the relationships between serum 25OHD levels and several clinical and laboratory parameters. P value will be considered significant if it was less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

Patients with SARS-CoV2 positive PCR

Exclusion Criteria:

Patients with chronic obstructive lung disease Chronic renal failure Patients with malabsorption Organ transplant recipient Pregnant women

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 100 patients who were diagnosed as SARS-CoV2 positive. The data will be collected from isolation hospital in Sohag governorate during the period from the start of June 2021 to the end of July 2021. Patients will be followed up for at least one month to evaluate the prognosis.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
serum level of vitamin D in patients who infected with COVID19 | during the period from the start of June 2021 to the end of July 2021

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Haridy, Deminstrator, Study Chair — Al-Azahar University; Mohamed Mahmoud, lecturer, Study Chair — Sohag University; Ahmed Nour-Eldin, lecturer, Study Chair — Sohag University; Asmaa Khalaf, lecturer, Study Chair — Sohag University; Amira Maher, lecturer, Study Chair — Sohag University
Locations (1):
- Mona Mohammed Abdelrahman, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masoud HH, Zaky S, Baki AA. Management Protocol for COVID-19 Patients Version 1.4/30th May 2020 Ministry of health and population (MOHP), Egypt. 2020;(September)
- [Background] Laird E, Rhodes J, Kenny RA. Vitamin D and Inflammation: Potential Implications for Severity of Covid-19. Ir Med J. 2020 May 7;113(5):81. PMID 32603576
- [Background] Mohammed M, Shafik NS, Maher A, Hemdan SB, Elhamed MA. Liver Injuries in COVID-19 infected patients. Sohag Medical Journal. 2020;24(2):15-19.